CLINICAL TRIAL: NCT02989870
Title: A Phase I Trial of Sorafenib and Bavituximab Plus Stereotactic Body Radiation Therapy (SBRT) for 1st Line Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: Sorafenib and Bavituximab Plus SBRT in Unresectable Hepatocellular Carcinoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No Interest. Investigator was unable to enroll any participants on study.
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18924
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: HepatoCellular Carcinoma; Unresectable HepatoCellular Carcinoma; Liver Cancer
Keywords: Liver Disease; Child-Pugh Class A; Child-Pugh Class B7
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Liver Diseases | interventions — Radiosurgery; Radiotherapy; Sorafenib; bavituximab; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SBRT, Sorafenib and Bavituximab (Experimental): This will be a 3+3 design with 3 dose cohorts. Following the dose escalation phase, an additional 6 patients will be enrolled as part of the dose expansion cohort.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT); Drug: Sorafenib; Drug: Bavituximab

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Participants will receive 3-5 fractions of radiation as determined by the dose level at time of enrollment. The starting dose level will be Dose Level 1: 8 Gy x 3 fractions for a total of 24 Gy. If sufficient treatment related toxicity is observed at the "initial starting dose", then the dose will be reduced to 16 Gy in 2 fractions of 8 Gy. The dose per fraction for each participant will be provided at the time of registration based on the toxicity experience of the previous participants on study. This will be escalated to 40 Gy in 5 fractions of 8 Gy.
  Other Names: radiotherapy
Drug: Sorafenib — Sorafenib by mouth (PO): 200 mg twice a day (BID) then 400 mg BID.
  Other Names: Nexavar; Kinase inhibitor
Drug: Bavituximab — Bavituximab intravenously (IV): 3 mg/kg every week (q wk).
  Other Names: Immunotherapy

SUMMARY:
This study involves a course of radiation to up to 5 tumors in the participant's liver followed by systemic therapy. (Treatment using substances that travel through the bloodstream, reaching and affecting cells all over the body.) The type of radiation is called stereotactic body radiation therapy (SBRT). The purpose of this study is to compare the effects, good and/or bad, of different doses of SBRT given along with the systemic therapies, sorafenib and bavituximab. The researchers want to see which dose of radiation will work best in stimulating the immune response and provide local control to the participant's liver. The usual treatment for hepatocellular carcinoma that is unresectable can be transarterial therapy, sorafenib alone and/or clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Advanced, unresectable hepatocellular carcinoma (unsuitable for resection, transplant or ablation)
* Age ≥ 18
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Must have normal organ and marrow function
* Childs-Pugh score of A or B7
* Must have measurable/evaluable disease as per RECIST 1.1 criteria
* Females of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential. For both males and females, effective methods of contraception must be used throughout the study and for four months following the last dose.
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Must be able to understand and be willing to sign the written informed consent form
* No more than 10 lesions in the liver

Exclusion Criteria:

* Have received radiation therapy, major surgery, other locoregional therapy, within 4 weeks prior to the first date of SBRT
* Prior radiotherapy to the region of the liver that would result in excessive doses to normal tissues due to overlap of radiation therapy fields
* Prior selective internal radiotherapy/hepatic arterial Yttrium therapy, at any time
* Any one hepatocellular carcinoma > 15 cm
* Total maximal sum of hepatocellular carcinomas or a single conglomerate HCC > 20 cm
* Direct tumor extension into the stomach, duodenum, small bowel or large bowel
* Measureable common or main branch biliary duct involvement with HCC
* Extrahepatic metastases or malignant nodes (that enhance with typical features of HCC) > 3.0 cm, in sum of maximal diameters (e.g., presence of one 3.4 cm metastatic lymph node or two 2 cm lung lesions). Note that benign non-enhancing periportal lymphadenopathy is not unusual in the presence of hepatitis and is permitted, even if the sum of enlarged nodes is > 2.0 cm.
* Use of regular phenytoin, carbamazepine, hypericum perforatum [also known as St. John's wort] or rifampin
* Have received sorafenib or other systemic therapies for treatment of HCC in the past.
* Active autoimmune disease; Patients with type I diabetes mellitus, hypothyroidism requiring only hormone replacement, psoriasis not requiring systemic treatment, or vitiligo are permitted for enrollment.
* No active malignancy except for nonmelanoma skin cancer or in situ cervical cancer. Patients surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before the trial are allowed.
* Myocardial infarction within past 6 months, congestive heart failure, unstable angina, active cardiomyopathy, unstable ventricular arrhythmia
* Congenital long QT syndrome
* Previous stroke within past 12 months
* Anti-coagulant therapy, bleeding or clotting disorder
* Symptomatic metastatic brain or meningeal tumors
* Presence of a non-healing wound, non-healing ulcer, or bone fracture
* History of organ allograft (including corneal transplant)
* Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial
* Women who are pregnant or breast-feeding
* Any condition which, in the investigator's opinion, makes the patient unsuitable for trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Occurrence of Treatment Related Adverse Events | From beginning of treatment to 30 days post-treatment, approximately 2 years
  Safety and tolerability, as assessed by presence of adverse events, serious adverse events, dose limiting toxicity (DLTs), abnormal laboratory parameters, vital signs. A DLT is defined as any toxicity not attributable to the disease or disease-related processes under investigation, which occurs from the start of radiation up to 42 days and is considered by the Investigators to be definitely, probably, or possibly related to the treatment. A DLT will be defined as any Grade 3 or higher treatment-related toxicity that occurs during the DLT evaluation period.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months post treatment
  Tumor response data will be summarized for dosed participants with measurable disease at baseline. Response will be evaluated using the international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. In addition, the immune response criteria will be utilized.
Progression Free Survival (PFS) | Up to 24 months post treatment
  PFS following SBRT, sorafenib, and bavituximab, will be summarized in the expansion phase arm. Progression will be evaluated using the international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression.) In addition, the immune response criteria will be utilized.
Overall Survival (OS) | Up to 24 months post treatment
  Overall Survival following SBRT, sorafenib, and bavituximab. OS: The length of time from beginning of study treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Frakes, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States